CLINICAL TRIAL: NCT03777540
Title: Post-Operative Outcomes And Predictors Of Mortality After Gastric Cancer Surgery In The Very Elderly Patients
Brief Title: Gastric Cancer Surgery in Elderly Patients
Acronym: GCSEP
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Marialuisa Lugaresi, Adjunct Professor, University of Bologna
Other Study IDs: Gastric Cancer Surgery
Record Dates: First submitted 2018-12-07; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age; timing of gastric resection: Patients 80-85 years; Patients > 85 years; Elective and urgent surgery.
  Interventions: Procedure: Gastric resection

INTERVENTIONS:
Procedure: Gastric resection — Partial gastrectomy with jejunal anastomosis," "total gastrectomy," "gastroenterostomy without gastrectomy" or "other" (palliative surgery).

SUMMARY:
Gastric cancer is most frequent after the fifth decade of life. Surgical risk is higher in aged population because of general health condition may affect the postoperative result. Aim of the study was to identify risk factors for post-operative mortality in octogenarian patients who underwent surgery for gastric cancer.

DETAILED DESCRIPTION:
236 patients (181: 80-85 years old and 55: >85 years old) underwent surgery for gastric cancer at the Sant'Orsola-Malpighi University Hospital in Bologna between 2010 and 2015. The variables of the two groups of patients were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed primary gastric cancer submitted to surgical treatment;
* Age > 80 years.

Exclusion Criteria:

* Patients with histologically confirmed primary gastric cancer submitted to surgical treatment and age < 80 years;
* Patients with histologically diagnosis of other neoplastic and non-neoplastic diseases submitted to surgical treatment.

Ages: 80 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 236 patients (181: 80-85 years old and 55: >85 years old) underwent surgery for gastric cancer at the Sant'Orsola-Malpighi University Hospital in Bologna between 2010 and 2015.
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Post-operative mortality In-hospital mortality was defined that occurred during hospitalization up to 90 days excluded post-operative mortality. Postoperative mortality | Up to 90-days
  mortality occurred up to 90 days from surgery

SECONDARY OUTCOMES:
Overall survival | Up to 5-years
  Overall survival was defined as the time from the date of surgery to patient death (including surgery-associated death or hospital death), or the date of last available information concerning vital status.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Nardo, MD,PhD, Study Chair — University of Bologna